CLINICAL TRIAL: NCT07389954
Title: Personalized Music Increases Dreaming During Propofol Sedation: A Randomized Trial Comparing Preferred Music, Matched Non-Preferred Music, and Silence
Brief Title: Personalized Music and Dreaming During Propofol Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wonkwang University Hospital (Other)
Responsible Party: Principal Investigator, Cheol Lee,MD,PhD,, Professor, Wonkwang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Wonkwang UH 24
Record Dates: First submitted 2026-01-19; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Conscious Sedation; Propofol; Dreams
Keywords: Procedural Sedation; Intravenous Sedation; Personalized Music; Preferred Music; Dream Recall; Dream Pleasantness

STUDY DESIGN:
Intervention Model Description: Single-center, parallel-group, three-arm randomized controlled trial. Participants were allocated 1:1:1 to Preferred Music, Matched Non-preferred Music, or Silence (headphones without playback) during IV propofol sedation.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Allocation was concealed and managed by a non-assessor audio technician. Standardized closed-back headphones were used in all arms (silence arm without playback). PACU interviewers, content coders, and statisticians were blinded to group assignment; scripted interactions and volume calibration supported blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Preferred Music (Experimental): Participants listen to their self-selected preferred music through standardized closed-back headphones during intravenous propofol sedation. Music starts at the beginning of sedation and continues until the end of the procedure/recovery period per protocol.
  Interventions: Behavioral: Preferred Music
- Matched Non-Preferred Music (Experimental): Participants listen to non-preferred music matched to the preferred-music selection (e.g., comparable tempo/energy/genre characteristics) through standardized closed-back headphones during intravenous propofol sedation. Playback timing and volume are standardized as in the preferred-music arm.
  Interventions: Behavioral: Matched Non-Preferred Music
- Silence (Headphones Only) (Placebo Comparator): Participants wear standardized closed-back headphones during intravenous propofol sedation, but no audio is played (silence condition). Procedures, timing, and staff interactions are otherwise identical to the music arms.
  Interventions: Behavioral: Silence (Headphones Only)

INTERVENTIONS:
Behavioral: Preferred Music — Standardized closed-back headphones are used to deliver music during IV propofol sedation. Depending on randomization, participants receive self-selected preferred music. Playback begins shortly before sedation and continues until the end of sedation; volume is calibrated per protocol.
  Arms: Preferred Music
Behavioral: Matched Non-Preferred Music — Standardized closed-back headphones are used to deliver music during IV propofol sedation. Depending on randomization, participants receive e matched non-preferred music. Playback begins shortly before sedation and continues until the end of sedation; volume is calibrated per protocol.
  Arms: Matched Non-Preferred Music
Behavioral: Silence (Headphones Only) — Participants wear identical closed-back headphones during IV propofol sedation, but no audio is played. Procedures, timing, and staff interactions are otherwise identical to the music arms.
  Arms: Silence (Headphones Only)

SUMMARY:
Many patients report dreams during intravenous (IV) propofol sedation, but it is uncertain whether listening to music changes how often dreams occur or how pleasant they feel. This single-center randomized study compared three auditory conditions during propofol sedation for elective surgery under spinal anesthesia or peripheral nerve block: (1) patient-selected preferred music, (2) matched non-preferred music, and (3) silence (headphones only). Music or silence was delivered through identical closed-back headphones starting 1-2 minutes before sedation and continuing until the end of sedation.

The main outcomes were (1) whether a dream occurred (yes/no) assessed by a neutral modified Brice interview in the post-anesthesia care unit (PACU), and (2) dream pleasantness rated on a 0-10 scale among participants who reported a dream. Additional outcomes included coded dream content features, patient satisfaction, sedative dose, hemodynamic variability, early recovery measures, postoperative symptoms, and adverse events.

DETAILED DESCRIPTION:
This is a single-center, parallel-group, three-arm randomized controlled trial evaluating the effects of auditory stimulation and music personalization on dreaming during IV propofol sedation. Adults (≥19 years) undergoing elective procedures under spinal anesthesia or peripheral nerve block with propofol sedation were eligible (ASA I-III). Participants were excluded for planned general anesthesia, severe hearing impairment, major psychiatric instability, expected significant bleeding, inability to complete interviews, or contraindication to sedative agents.

Randomization and blinding: Participants were randomized 1:1:1 to Preferred Music, Matched Non-preferred Music, or Silence using computerized randomization with variable block sizes, stratified by procedure category and preoperative anxiety (STAI-State tertiles). Allocation was concealed. An audio technician (non-assessor) set up the assigned condition. PACU interviewers, dream-content coders, and statisticians were blinded. Standardized closed-back headphones were used for all groups, with scripted staff interactions and calibrated volume (50-60 dB(A)) to support blinding; blinding integrity was assessed by questionnaire.

Interventions:

• Preferred Music: Participants selected one personally meaningful track preoperatively. The track was played continuously on loop through closed-back headphones starting 1-2 minutes before sedative infusion and continued until the end of sedation.

Final-The effect of Auditory St…

* Matched Non-preferred Music: Participants listened to a pleasant non-selected track matched to the preferred selection for tempo (±10 bpm), genre family, and loudness to separate preference effects from acoustic features; playback timing was identical.
* Silence Control: Participants wore identical headphones for the same duration without audio playback.

Sedation protocol and monitoring: Propofol was administered per a standardized regimen (initial bolus 0.5-1 mg/kg followed by infusion 25-75 µg/kg/min) titrated to maintain BIS 65-85. Sedation depth was assessed using MOAA/S (primary) and RASS (secondary), with routine physiologic monitoring and supplemental oxygen.

Outcomes: Co-primary outcomes were (1) dream incidence (yes/no) assessed by a neutral modified Brice interview in PACU, with the primary contrast of Music-pooled (Preferred or Non-preferred) versus Silence; and (2) dream pleasantness (0-10 numeric scale) among recallers, with the primary contrast of Preferred versus Matched Non-preferred music. PACU interview timing used prespecified readiness criteria and was initiated at approximately 15 minutes (±5) after PACU arrival, repeated every 5-10 minutes if needed up to 60 minutes. Secondary outcomes included blinded coded dream content features, patient satisfaction, sedative dose, hemodynamic variability, recovery endpoints (e.g., Aldrete-based recovery and PACU length of stay), postoperative symptoms (pain, nausea/vomiting, shivering), and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ [19] years and ≤ [70] years.
* Scheduled for an elective procedure under intravenous propofol sedation at Wonkwang University Hospital.
* American Society of Anesthesiologists (ASA) physical status I-III.
* Able to understand the study procedures and provide written informed consent.

Exclusion Criteria:

* Known hearing impairment that would interfere with headphone-based auditory intervention.
* Pre-existing cognitive impairment or delirium at baseline (e.g., diagnosed dementia or active delirium).
* Use of sedatives, hypnotics, or psychoactive medications that could confound dreaming assessment, per protocol.
* Significant neurologic or psychiatric disorder that may affect dream recall/reporting.
* Inability to complete the postoperative PACU interview or inability to communicate reliably.
* Any condition judged by the investigator to make participation unsafe or data uninterpretable.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2025-12-19 (Actual); Primary Completion 2026-01-16 (Actual); Study Completion 2026-01-16 (Actual)

PRIMARY OUTCOMES:
Dream Incidence (Yes/No) by Modified Brice Interview | PACU: primary at 15 minutes (±5) after arrival; if not ready, repeated every 5-10 minutes up to 60 minutes (first valid interview within 60 minutes).
  Dream occurrence (yes/no) assessed using a neutral modified Brice interview during early recovery in the PACU. Primary comparison: Music-pooled (Preferred or Non-preferred) vs Silence.
Dream Pleasantness (0-10 Numeric Rating Scale) Among Recallers | Same PACU interview window as above: 15 minutes (±5) after PACU arrival; repeated every 5-10 minutes up to 60 minutes until readiness is met (first valid interview within 60 minutes).
  Dream pleasantness rated on a 0-10 Dream Pleasantness Numeric Rating Scale (minimum 0, maximum 10), where higher scores indicate more pleasant dreams (0 = not pleasant at all, 10 = extremely pleasant).

SECONDARY OUTCOMES:
Dream Content Metrics (Blinded Coding) Among Recallers | PACU interview window: first valid interview within 60 minutes after PACU arrival.
  Among participants with dream recall, dream content is assessed using prespecified blinded coding. Metrics include: (a) music-thematic incorporation (present/absent); (b) auditory salience score (0-3; 0 = none, 3 = strong; higher scores indicate greater auditory incorporation); (c) affect valence score (-2 to +2; -2 = very negative, +2 = very positive; higher scores indicate more positive affect); (d) vividness score (0-10; 0 = not vivid, 10 = extremely vivid; higher scores indicate more vivid dreams); and (e) sense of control/agency score (0-10; 0 = no control, 10 = complete control; higher scores indicate greater perceived control/agency). Narratives are double-coded with adjudication for disagreements.
Patient Satisfaction (1-5 Scale) | PACU (early recovery; within the PACU assessment period).
  Patient satisfaction is assessed during early recovery in the PACU using a 5-point Likert satisfaction scale (minimum 1, maximum 5), where higher scores indicate greater satisfaction (1 = very dissatisfied, 5 = very satisfied).
Intraoperative Mean Arterial Pressure Variability (Standard Deviation) | During sedation (intraoperative period).
  Variability in mean arterial pressure (MAP) is quantified as the standard deviation (SD) of continuously recorded MAP values during the propofol sedation period. Unit: mmHg. Higher SD indicates greater blood pressure variability. as standard deviation during the sedation period.
Intraoperative Heart Rate Variability (Standard Deviation) | During sedation (intraoperative period).
  Variability in heart rate (HR) is quantified as the standard deviation (SD) of continuously recorded HR values during the propofol sedation period. Unit: beats per minute (bpm). Higher SD indicates greater heart rate variability.
Total Propofol Dose Administered | During procedure and immediate recovery period.
  Total propofol administered during the procedure is recorded. Dose is expressed as mg/kg (weight-adjusted total dose). Higher values indicate greater propofol exposure.
Total Opioid Consumption (Morphine Milligram Equivalents) | During procedure and immediate recovery period.
  Total opioid consumption during the procedure and immediate recovery is converted to morphine milligram equivalents (MME) and recorded in mg. Higher values indicate greater opioid exposure
Vasopressor Use (Yes/No) | During procedure and immediate recovery period.
  Any vasopressor administration during the procedure and immediate recovery is recorded as yes/no. Higher values (yes) indicate that vasopressor support was required.
Time to Recovery (Aldrete Score ≥ 9) and PACU Length of Stay | From PACU arrival until discharge criteria met / PACU discharge.
  Time to achieve Aldrete score ≥9 and total PACU time (minutes).
Postoperative Pain Intensity (0-10 Numeric Rating Scale) | PACU stay (early recovery).
  Postoperative pain intensity is assessed during early recovery in the PACU using a 0-10 Numeric Rating Scale (NRS; minimum 0, maximum 10), where higher scores indicate worse pain (0 = no pain, 10 = worst imaginable pain).
Postoperative Nausea and Vomiting Severity (0-3 Ordinal Scale) | PACU stay (early recovery).
  Postoperative nausea and vomiting (PONV) severity is assessed during early recovery in the PACU using a 0-3 ordinal PONV severity scale (minimum 0, maximum 3), where higher scores indicate worse symptoms (0 = none, 1 = mild nausea, 2 = moderate/severe nausea or retching, 3 = vomiting).
Postoperative Shivering (Yes/No) | PACU stay (early recovery).
  Postoperative shivering during early recovery in the PACU is recorded as present/absent (yes/no).
Unplanned Hospital Admission (Yes/No) | From procedure start through PACU discharge.
  Any unplanned hospital admission from procedure start through PACU discharge is recorded as yes/no (higher = yes indicates admission occurred).
dverse Events (Number of Events) | From procedure start through PACU discharge.
  The total number of adverse events occurring from procedure start through PACU discharge is recorded per protocol (higher values indicate more events).
Any Adverse Event (Yes/No) | From procedure start through PACU discharge.
  Occurrence of any adverse event from procedure start through PACU discharge is recorded as yes/no (higher = yes indicates an event occurred).

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Lee, M.D.,Ph.D, Principal Investigator — Department of anesthesiology and pain medicine, Wonkwang University Hospital
Locations (1):
- IRB of Wonkwnag University Hospital, Iksan, South Korea